CLINICAL TRIAL: NCT03071978
Title: Application of Right Atrial Left Ventricular Fusion Pacing in Patients With CRT (Cardiac Resynchronization Therapy) Indications
Brief Title: Application of Right Atrial Left Ventricular Fusion Pacing in Patients With CRT Indications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LV Study
Record Dates: First submitted 2017-01-23; First posted 2017-03-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; LV-fusion pacing; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LV-fusion pacing (Experimental): Left Ventricular pacing (without Right Ventricular pacing)
  Interventions: Device: CRT with LV-only pacing / bi-ventricular pacing
- BV pacing (Active Comparator): Bi-Ventricular pacing
  Interventions: Device: CRT with LV-only pacing / bi-ventricular pacing

INTERVENTIONS:
Device: CRT with LV-only pacing / bi-ventricular pacing — LV-fusion pacing group received cardiac resynchronization therapy with adaptive algorithm and disabled RV pacing. While BV pacing group received conventional cardiac resynchronization therapy without adaptive algorithm.

SUMMARY:
This study is designed to assess the clinical outcomes of Left-Ventricular (LV) fusion pacing compared to Bi-Ventricular (BV) pacing, also known as Cardiac Resynchronization Therapy (CRT), in Chinese Heart Failure (HF) population. Specifically, the study will assess the changes of cardiac function of each group through 3-month follow up/ 6-month follow up compared with original outcomes before aCRT (adaptive Cardiac Resynchronization Therapy) implantation. Secondly, the study will assess whether parameters of aCRT that were tested in Western population are relevant to parameters of Chinese HF patients.

DETAILED DESCRIPTION:
Traditional dual-chamber pacemakers usually utilize pacing at right atrium (RA) and right ventricle (RV). But many clinical studies have proved that permanent RV pacing could cause ventricular desynchronization in electrical activation and mechanical movement, also may lead to atrial fibrillation and cardiac failure in the long term. Cardiac Resynchronization Therapy (CRT) can overcome the ventricular desynchrony caused by permanent RV pacing, through pacing both left and right ventricles. But the cost of CRT device is usually expensive in emerging markets like in China. Recently, a few clinical studies have demonstrated that LV-fusion pacing (without RV pacing) using adaptive CRT feature provides better clinical outcomes than RV pacing, and also equivalent clinical improvements compared to conventional CRT pacing. However, it is unknown whether similar results can be duplicated in Chinese population as the clinical profile of Chinese CRT populations is different from that of Western CRT population.

This study is designed to assess the clinical outcomes of Left-Ventricular (LV) fusion pacing compared to Bi-Ventricular (BV) pacing in Chinese Heart Failure population. Specifically, the study will assess the changes of cardiac function of each group through 3-month follow up/ 6-month follow up compared with original outcomes before aCRT implantation. Secondly, the study will assess whether parameters of aCRT that were tested in Western population are relevant to parameters of Chinese HF patients.

CRT-indicated heart failure patients who meet the Inclusion & Exclusion criteria will be enrolled voluntarily in this study. No intervention will be assigned to enrolled patients. CRT therapy will be assigned according to the Guideline (ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012). Left-Ventricular (LV) fusion pacing or Bi-Ventricular (BV) pacing mode, both included in CRT therapy, will be applied upon physicians' judgment based on the Guideline and patients' specific situations. Both pacing modes, as well as all the clinical assessments in this study, are routine cares in clinical practice.

The study will enroll up to 30 subjects in each group (LV pacing group and BV pacing group) that meet the indication for CRT therapy, and also the Inclusion & Exclusion criteria. Consented subjects will receive CRT therapy and two follow-ups in the following 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18~80
* Life expectancy > 1 year
* Sign Informed Consent
* CRT-indicated
* NYHA (New York Heart Association) class II and III
* PR (term in Electrocardiograph) interval < 200 ms
* ECG (Electrocardiograph) LBBB (left bundle branch block)

Exclusion Criteria:

* Patient with severe liver or kidney dysfunction
* CRT-contraindication
* CRT-upgraded
* Persistent AF (atrial fibrillation)
* AV block (atrioventricular block)
* RBBB (right bundle branch block)
* Valvular Disease
* LV threshold ≥ 3.5 volt
* Patient is unwilling to sign the informed consent
* Patient is pregnant or has pregnancy intention in the study duration
* Patient has a medical condition that would limit study participation
* Patient is enrolled in a concurrent study that may affect the outcome of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) | 6-month follow up after CRT implantation
  Change of Left Ventricular Ejection Fraction (LVEF) from Baseline to 6-month follow-up

SECONDARY OUTCOMES:
New York Heart Association (NYHA) class | 6-month follow up after CRT implantation
  Change of New York Heart Association (NYHA) class from Baseline to 6-month follow-up
6-minute walking distance (6MWD) | 6-month follow up after CRT implantation
  Change of 6-minute walking distance (6MWD) from Baseline to 6-month follow-up
ECG QRS duration | 6-month follow up after CRT implantation
  Change of ECG QRS duration from Baseline to 6-month follow-up
echocardiographic assessments (including LVESV, LVEDV, LVESD, LVEDD) | 6-month follow up after CRT implantation
  Change of echocardiographic assessments (including LVESV, LVEDV, LVESD, LVEDD) from Baseline to 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yan-gang Su, M.D., Principal Investigator — ZhongShan Hospital, Shanghai; Shu Zhang, M.D., Principal Investigator — Fuwai Hospital, Beijing
Locations (5):
- China (5):
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Greentown Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No